CLINICAL TRIAL: NCT01746407
Title: Observational Study to Procure Human Specimens for Use in the Diagnosis and Management of Sepsis and Other Related Conditions
Brief Title: Procurement of Human Specimens for the Evaluation of Early Markers of Sepsis
Acronym: EMOS
Status: Completed | Type: Observational
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Other Study IDs: 09DELK12
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Infection
Keywords: Emergency Department; Infection; Sepsis
MeSH Terms: conditions — Infections; Emergencies; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples stored @ -70C.
Oversight: Data Monitoring Committee: No

SUMMARY:
Procure blood specimens from individuals presenting to the emergency department (ED) with signs and /or symptoms of systemic infection or sepsis. The samples will be used for research and development activities related to sepsis, infections, etc.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age or older
* For women of child bearing years: not known to be pregnant
* Blood culture ordered as part of the ED, ICU (or equivalent) or hospital floor stay.

Exclusion Criteria:

* Previously enrolled in this study
* Vulnerable individual
* Unable to speak and/or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presentation to an emergency department
Sampling Method: Non-Probability Sample
Enrollment: 872 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression of infection to severe sepsis | 72 hours
  Assessment of the progression of infection to severe sepsis in an ED population who present with signs or symptoms of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Greg S Martin, MD, M.Sc., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia